CLINICAL TRIAL: NCT00974987
Title: A Phase II, Multicenter, Study for Newly Diagnosed Glioblastomas Using Boron Neutron Capture Therapy, Additional X-ray Treatment and Chemotherapy
Brief Title: Boron Neutron Capture Therapy, Radiation Therapy, and Temozolomide in Treating Patients With Newly Diagnosed Glioblastoma Multiforme
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Translational Research Center for Medical Innovation, Kobe, Hyogo, Japan (Other)
Collaborators: Department of Nuerosurgery, Osaka Medical College (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSAKA-TRIBRAIN0902; CDR0000650829 (Registry Identifier: PDQ (Physician Data Query)); UMIN000002385 (Registry Identifier: UMIN CTR)
Record Dates: First submitted 2009-09-10; First posted 2009-09-11 (Estimated); Last update posted 2018-04-25 (Actual); Status verified 2017-06

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult giant cell glioblastoma; adult glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Gliosarcoma | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment group (Experimental): BNCT(boron neutron capture therapy), XRT(X-ray radiation treatment) and TMZ(temozolomide) treatment
  Interventions: Radiation: BNCT(boron neutron capture therapy); Radiation: XRT(X-ray radiation treatment); Drug: TMZ(temozolomide)

INTERVENTIONS:
Radiation: BNCT(boron neutron capture therapy) — BSH(sodium borocaptate) 100mg/kg iv for one hour starting 13 hours before irradiation, and BPA(p-boronophenylalanine) 500/mg/kg iv at a speed of 200mg/kg/hr for 2 hours starting 2 hours before irradiation. During irradiation, BPA iv continues at a speed of 100mg/kg/hr.
Radiation: XRT(X-ray radiation treatment) — After BNCT, 2Gy irradiation every day for 12 days.
Drug: TMZ(temozolomide) — 75mg/m2 for day1-12. After XRT, repeat the cycle of 150-200mg/m2 for 5 days and cessation for 23 days.

SUMMARY:
RATIONALE: Boron neutron capture therapy and radiation therapy use high-energy x-rays and other types of radiation to kill tumor cells. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving boron neutron capture therapy followed by radiation therapy and temozolomide may kill more tumor cells.

PURPOSE: This phase II trial is studying the side effects of giving boron neutron capture therapy together with radiation therapy and temozolomide in treating patients with newly diagnosed glioblastoma multiforme.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate the overall survival of patients with newly diagnosed glioblastoma multiforme treated with boron neutron capture therapy, radiotherapy, and concurrent and adjuvant temozolomide.
* Evaluate tumor response in patients treated with this regimen.
* Evaluate the adverse effects of this regimen in these patients.

OUTLINE: This is a multicenter study.

Patients undergo boron neutron capture therapy followed by radiotherapy and concurrent and adjuvant oral temozolomide.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed glioblastoma multiforme

  * Newly diagnosed disease
* Tumor located at a supratentorial hemisphere

  * Deepest part of tumor < 6 cm from the scalp
  * Bottom of the tumor > 6 cm from the scalp allowed provided air instillation into tumor-removed cavity is possible
* No cerebrospinal fluid dissemination

PATIENT CHARACTERISTICS:

* Karnofsky performance status 70-100%
* Life expectancy > 3 months
* Leukocyte count ≥ 3,000/μL
* Platelet count ≥ 10.0 × 10^4/μL
* Hemoglobin ≥ 8.0 g/dL
* Serum creatinine ≤ 1.5 mg/dL
* ALT and AST ≤ 100 IU/L
* No phenylketonuria
* Not pregnant or nursing
* No NYHA class III-IV heart failure
* No patient whose participation in the present study is considered inappropriate by a Principal Investigator or Clinical Investigator

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy or radiotherapy

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2009-09-01 (Actual); Primary Completion 2016-02-29 (Actual); Study Completion 2016-02-29 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) | Time to death from BSH injection（up to 6 years）

SECONDARY OUTCOMES:
Tumor response（RECIST） | From BSH injection to the end of treatment, whichever came first, assessed up to 96 weeks
Objective Response Rate (ORR) | From BSH injection to the end of treatment, whichever came first, assessed up to 96 weeks
Disease Control Rate (DCR) | From BSH injection to the end of treatment, whichever came first, assessed up to 96 weeks
Adverse event | Time to final follow-up survey from the date of enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Shin-Ichi Miyatake, MD, PhD, Principal Investigator — Osaka Medical College
Locations (1):
- Osaka Medical College, Takatsuki, Osaka, Japan

REFERENCES:
- [Result] Kawabata S, Miyatake S, Hiramatsu R, Hirota Y, Miyata S, Takekita Y, Kuroiwa T, Kirihata M, Sakurai Y, Maruhashi A, Ono K. Phase II clinical study of boron neutron capture therapy combined with X-ray radiotherapy/temozolomide in patients with newly diagnosed glioblastoma multiforme--study design and current status report. Appl Radiat Isot. 2011 Dec;69(12):1796-9. doi: 10.1016/j.apradiso.2011.03.014. Epub 2011 Mar 21. PMID 21459588